CLINICAL TRIAL: NCT01917344
Title: The Brain, Neurological Features and Neuropsychological Functioning in Adults With Phenylketonuria: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Susan Waisbren, Susan Waisbren, P.h.D, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-P00003864
Record Dates: First submitted 2013-08-05; First posted 2013-08-06 (Estimated); Results first posted 2015-06-19 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-06

CONDITIONS: Phenylketonuria
Keywords: Phenylketonuria; MRI; Neuropsychological functioning; Neurological functioning; EEG
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adults with PKU (Other): MRI, EEG, neuropsychological testing, neurological examination, blood draw, diet diary, physical examination. These activities were performed for the study, but no drug or other interventions took place.
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI

SUMMARY:
Newborn screening and early treatment prevent the most severe manifestations of phenylketonuria (PKU). However, executive functioning deficits, attention deficit disorder, slow processing speed, and visual-motor problems commonly occur. Many adults with this disorder also suffer depression and anxiety. Using advanced electroencephalogram (EEG) and magnetic resonance imaging (MRI) techniques, including novel MR spectroscopy (MRS) we hope to discover why this distinct constellation of deficits occurs in PKU. Adult subjects with PKU will undergo EEG and comprehensive MRI evaluations, including a novel method of MR spectroscopy to determine brain phenylalanine levels. In addition, they will receive neurological and neuropsychological examinations and dietary evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Adult with classic PKU who has been seen at one of the hospitals collaborating in this study
2. Age 18-55 years
3. Medical Records available that include genotype and blood phenylalanine levels during the first 6 years of life. (We have over 300 patients with PKU with genotypes in our clinic, of whom about half are adults.)
4. Capable of providing informed consent
5. Able to undergo MRI procedures without sedating medication
6. Does not have metal implants
7. Not currently on Kuvan, Large Neutral Amino Acid therapy or involved in any clinical trials.

   -

Exclusion Criteria:

1. Mild PKU or mild hyperphenylalaninemia
2. Less than 18 years old or great than 55 years old
3. No medical records available for the first 6 years of life
4. No record of genotype
5. Not capable of providing informed consent
6. Not able to undergo MRI without sedating medication
7. Has metal implants
8. Currently taking Kuvan, Large Neutral Amino Acid therapy or involved in any clinical trial

   -

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2013-08; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan E Waisbren, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A recruitment letter was sent to adults with PKU who were not enrolled in another clinical trial.
Groups:
- Adults With PKU: MRI, EEG, neuropsychological testing, neurological examination, blood draw, diet diary, physical examination
  MRI
Period: Overall Study
Arm/Group | Adults With PKU
Started | 10
Completed | 9
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Adults (ages 18 and older) with phenylketonuria (PKU)
Arm/Group | Adults With PKU
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants] — Brain and Blood Phenylalanine
  Participants
    <=18 years | 0
    Between 18 and 65 years | 10
    >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Phenylalanine Level in the Brain as Determined by MR Spectroscopy and in Blood
Description: Brain Phe levels (umol/L) using MRI correlated spectroscopy and Blood Phe levels (umol/L) obtained on the same day.
Time Frame: During period of evaluation, approximately 8 hours
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Adults With PKU
Number analyzed (Participants) | 9
umol/L
  White Matter | 130 (38)
  Gray Matter | 137 (24)
  Blood Phe level | 961 (378)

2. Secondary Outcome: Full Scale Intelligence Quotient (IQ)
Time Frame: During period of evaluation, approximately 8 hours
Reporting Status: Not Posted

3. Secondary Outcome: Electroencephalogram (EEG) Findings
Time Frame: During period of evaluation, approximately 8 hours
Reporting Status: Not Posted

4. Secondary Outcome: Volumetric MRI Findings
Time Frame: During period of evaluation, approximately 8 hours
Reporting Status: Not Posted

5. Secondary Outcome: Diffusion Tensor Imaging (DTI) Findings Through MRI
Time Frame: During period of evaluation, approximately 8 hours
Reporting Status: Not Posted

6. Secondary Outcome: Tremor as Determined Through Neurological Evaluation
Time Frame: During period of evaluation, approximately 8 hours
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Two years.
Arm/Group | Adults With PKU
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes